CLINICAL TRIAL: NCT07399496
Title: Accelerated Transcranial Magnetic Stimulation (TMS) for Apathy in Parkinson's Disease
Brief Title: Accelerated TMS for Apathy in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Daniel Lench, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00147039
Record Dates: First submitted 2026-01-07; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: Neuromodulation; iTBS; Transcranial Magnetic Stimulation; Apathy; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS group (Other): participants with Parkinson's disease and clinically significant apathy receive accelerated iTBS rTMS targeting the left dorsomedial prefrontal cortex (dmPFC) using a MagVenture MagPro system with a cooled figure-of-eight coil and Brainsight neuronavigation (slightly off midline). Resting motor threshold (rMT) is determined on the first stimulation visit (PEST) and stimulation is delivered at 120% rMT. Treatment occurs on 6 days over ~2 weeks (days may be non-contiguous), with 8 sessions/day separated by 10-15 min. Each session delivers 600 pulses (50 Hz triplets; 2 s on/8 s off; ~190 s), totaling 4,800 pulses/day and 28,800 pulses overall. Coil position/angle and scalp-to-cortex distance are tracked; tolerability/acceptability (headache, pain, scalp irritation, facial twitching, fatigue, fear/anxiety) is assessed before/after sessions.
  Interventions: Device: Accelerated intermittent theta-burst stimulation (iTBS) rTMS to left dorsomedial prefrontal cortex (dmPFC)

INTERVENTIONS:
Device: Accelerated intermittent theta-burst stimulation (iTBS) rTMS to left dorsomedial prefrontal cortex (dmPFC) — Accelerated intermittent theta-burst stimulation (iTBS) rTMS to left dorsomedial prefrontal cortex (dmPFC) (MagVenture MagPro with cooled figure-of-eight coil; Brainsight neuronavigation; 120% rMT; 6 treatment days over ~2 weeks; 8 sessions/day; 600 pulses/session; 10-15 min inter-session interval).

SUMMARY:
This single-site, open-label pilot study will evaluate the feasibility, tolerability, and preliminary efficacy of accelerated intermittent theta-burst stimulation (iTBS) targeting the dorsomedial prefrontal cortex (dmPFC) for apathy in individuals with Parkinson's Disease (PD). Fifteen participants with PD and clinically significant apathy will undergo six treatment visits over two weeks, receiving eight iTBS sessions per day. Outcomes include adherence, tolerability, changes in apathy (Lille Apathy Rating Scale), functional engagement, and neural target engagement assessed via resting-state fMRI and EEG. Follow-up assessments will occur at two and four weeks post-treatment.

DETAILED DESCRIPTION:
This study is designed to explore a new treatment option for people with Parkinson's disease who experience apathy, which means loss of motivation or interest in daily activities. Apathy is common in Parkinson's disease and can lower quality of life, but current treatments are limited. Investigators are testing whether a non-invasive brain stimulation technique called repetitive transcranial magnetic stimulation (rTMS) is tolerable, acceptable and can be used to improve apathy in patients with Parkinson's disease. TMS delivers brief magnetic pulses to specific areas of the brain that are linked to motivation and decision-making. In this study, Investigators will use an "accelerated" version of TMS, which gives several short sessions in a single day, reducing the number of visits required. The purpose of this research is to see whether this treatment approach is feasible, tolerable and and potentially effective at treating apathy in people with Parkinson's disease. If successful, this research study will hopefully lead to a larger study in the future where the efficacy of the treatments can be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-85
* Diagnosis of Parkinson's Disease
* AES ≥37
* Stable PD medications
* Caregiver informant available

Exclusion Criteria:

* MRI/TMS contraindications
* Severe cognitive impairment (MoCA <21)
* Psychiatric disorders (bipolar, schizophrenia, PTSD)
* Seizure history
* Pregnancy

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
TMS adherence | Day 1 through Day 14 (6 treatment days over approximately 2 weeks)
  Proportion of planned accelerated iTBS sessions completed. Adherence is calculated as number of iTBS sessions completed out of 48 scheduled sessions (6 treatment days × 8 sessions/day).
TMS tolerability and acceptability | Measured during each treatment day (6 days within a 2-week period)
  Participant-reported tolerability/acceptability assessed with a standardized questionnaire capturing frequency and severity of common TMS side effects (e.g., headache, pain, scalp irritation, facial twitching, fatigue, fear/anxiety), collected during treatment days (pre/post sessions).
Apathy severity | Baseline (Day 0), immediately post-treatment (Day 14), 2 weeks post-treatment, and 4 weeks post-treatment
  Change in apathy measured by the Lille Apathy Rating Scale (LARS) patient and caregiver/informant versions; analyzed as change from baseline to post-treatment and follow-up timepoints.
Target engagement (dmPFC network modulation) | Baseline MRI/EEG assessments (Days 0-1) and post-treatment MRI/EEG assessments (Days 14-15)
  Change in dmPFC target engagement measured by (1) resting-state fMRI functional connectivity of dmPFC to motivation/effort-related nodes and (2) EEG waveform/response metrics during motivation/effort tasks, comparing pre- vs post-intervention.

SECONDARY OUTCOMES:
Goal attainment | Baseline (Day 0), immediately post-treatment (Day 14), 2 weeks post-treatment, and 4 weeks post-treatment
  Change in goal-directed behavior measured by Bangor Goal-Setting Interview outcomes, including proportion/percent attainment of individualized goals across assessment timepoints.
Change in apathy as measured by the Dimensional Apathy Scale | Baseline (Day 0), immediately post-treatment (Day 14), 2 weeks post-treatment, and 4 weeks post-treatment"
  Change in apathy-related symptoms measured using the Dimensional Apathy Scale (DAS), including patient/informant reports where applicable.
Change in apathy-related behavior as measured by the Frontal Systems Behavior Scale | Baseline (Day 0), immediately post-treatment (Day 14), 2 weeks post-treatment, and 4 weeks post-treatment"
  Change in apathy-related symptoms measured using the Frontal Systems Behavior Scale (FRSBE), including patient/informant reports where applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lench, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States